CLINICAL TRIAL: NCT00849238
Title: Mycophenolate Mofetil Maintenance Therapy for Liver Transplantation Following Campath-1H Induction
Brief Title: Mycophenolate Mofetil Maintenance Therapy for Liver Transplantation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: feasibility issues
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: H-2005-0291; CEL
Record Dates: First submitted 2007-12-14; First posted 2009-02-23 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Primary Liver Transplant
MeSH Terms: interventions — Mycophenolic Acid

INTERVENTIONS:
Drug: mycophenolate mofetil

SUMMARY:
The rationale for this study is to determine if Campath-1H can be used in liver transplant recipients to induce a state of immunological unresponsiveness that would not only eliminate the need for calcineurin inhibitors maintenance therapy, but also reduce corticosteroids utilization, decreasing the incidence of acute cellular rejection and perhaps reduce the severity of histologic recurrence of certain autoimmune diseases responsible for causing liver failure. The investigator propose a randomized prospective open label trial in 50 liver transplant recipients who will received a calcineurin inhibitors free immunosuppressive protocol that consist of a single dose of Campath-1H as an induction therapy in association with maintenance mycophenolate mofetil (CellCept®) and low dose steroids. The second group will receive a standard immunosuppressive regimen, which consists of IV steroid induction therapy and maintenance steroids, together with tacrolimus at a full therapeutic dose with no induction antibody therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects;
2. Ages 45 years and older;
3. Are to receive a liver transplant.

Exclusion Criteria:

1. Recipients of a multi-organ transplant;
2. known hypersensitivity to daclizumab, CellCept®, or prednisone;
3. therapy with an investigational medication within 4 weeks of study entry;
4. history of malignancies within the past 5 years and/or lymphoma, excluding adequately treated skin carcinoma (basal or squamous cell), or other than exclusion #9;
5. history of a psychological illness or condition such as to interfere with the patient's ability to understand the requirements of the study;
6. history of HIV infection;
7. females who are pregnant or nursing;
8. subject is receiving systemic corticosteroids for other medical conditions for which the physician feels that discontinuation of corticosteroids is contraindicated;
9. T2 or higher hepatocellular carcinoma

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)